CLINICAL TRIAL: NCT01013129
Title: Genetic Susceptibility, Environment & Prostate Cancer Risk
Brief Title: Studying Genes, Environment, and Prostate Cancer Risk in Patients With or Without Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Portland VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jackilen Shannon, Staff Scientist, Portland VA Medical Center
Other Study IDs: CDR0000648179; VAMC-OR-M1736; CPC-07129-L
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Hereditary Prostate Cancer; Prostate Cancer
Keywords: hereditary prostate cancer; prostate cancer
MeSH Terms: conditions — Prostate cancer, familial; Prostatic Neoplasms | interventions — Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10ml blood specimen drawn from probands consented in person at the Portland VA; saliva samples from all consented probands (N = 748).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Probands
  Interventions: Genetic: DNA analysis; Genetic: polymorphism analysis; Other: laboratory biomarker analysis; Other: medical chart review; Other: questionnaire administration; Procedure: evaluation of cancer risk factors; Procedure: study of high risk factors

INTERVENTIONS:
Genetic: DNA analysis — saliva samples will be collected from men (probands) who join the study.
Genetic: polymorphism analysis — we will genotype DNA samples (buccal) from all probands and conduct a traditional case-control analysis
Other: laboratory biomarker analysis — 10ml blood specimen will be obtained and processed (on probands locally-consented and/or those who have an appointment at the VA in Portland, Oregon) to allow for analyses of erythrocyte fatty acids and future nutrient and DNA analyses
Other: medical chart review — PSA results, prostate biopsy pathology reports and clinician notes related to the biopsy are reviewed for final data analysis
Other: questionnaire administration — probands are asked to complete questionnaires on 1) family history of cancer, 2) diet history over the past year, 3) employment environment and risk factors and/or 4) changes to diet, medications since enrollment in originating case control study
Procedure: evaluation of cancer risk factors — pathology reports will be reviewed for probands whose prostate biopsies reveal cancer; these factors will be evaluated for cancer risk factors
Procedure: study of high risk factors — prostate biopsy pathology reports will be reviewed for high risk factors

SUMMARY:
RATIONALE: Gathering information about genetic and environmental factors may help doctors learn more about a person's risk for developing prostate cancer.

PURPOSE: This research project is studying genes, environment, and prostate cancer risk in patients with or without prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the association between variation in genes involved in ROS detoxification, oxidative stress response, and prostate cancer risk.
* To determine the association between fatty acid levels and prostate cancer risk.

OUTLINE: Probands undergo blood and saliva sample collection for fatty acid, DNA, and polymorphism analyses. Archived blood and tissue samples from probands who previously participated in Dr. Shannon's Diet and Prostate Cancer Risk study are also analyzed. Medical records of probands are reviewed for demographics, history and course of disease, and clinical laboratory test results.

All probands completed the "Genetic Risk Easy Assessment Tool Family History of Cancer" and "Diet History and Environmental Risk Factor" questionnaires at baseline. If a proband previously participated on our Diet and Prostate Cancer Risk study, he was asked to complete the "Changes in Diet, Prescriptions, Supplementals and Herbal Remedies" questionnaire in addition to the "Genetic Risk Easy Assessment Tool Family History of Cancer" questionnaire at baseline for this study.

PROJECTED ACCRUAL: A total of 750 participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Prior diagnosis of prostate cancer or negative prostate biopsy AND previously participated in Dr. Shannon's Diet and Prostate Cancer Risk study and consented to future studies (proband)
  * Referred to the Portland VA Medical Center urology clinic for a prostate biopsy (proband)

    * Introduced to this study by a proband OR found to be related to a proband who is part of a homogenous high-risk subgroup after completion of the family history of cancer analysis

PATIENT CHARACTERISTICS:

* See Disease Characteristics

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 21 Years to 120 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Recontacting previously recruited Diet and Prostate Cancer Risk study participants; cases and biopsy negative controls
  2. Prospective recruitment of men referred for a prostate biopsy to the Portland VA urology clinic
  3. Men from the public sector who learn about our study and would like to participate
Sampling Method: Non-Probability Sample
Enrollment: 748 (Actual)
Dates: Start 2008-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Association between variation in genes involved in reactive oxygen species detoxification, oxidative stress response, and prostate cancer risk | through study completion; 1 day
  Using saliva samples, we conducted analysis on probands' oxidative stress pathway genes and whether these were associated with prostate cancer risk.
Association between blood fatty acids and prostate cancer risk | through study completion; 1 day
  Using blood samples, we conducted analysis on probands' fatty acid level and whether these were associated with prostate cancer risk.

CONTACTS AND LOCATIONS:
Overall Officials: Jackilen Shannon, PhD, Principal Investigator — Portland VA Medical Center
Locations (1):
- Veterans Affairs Medical Center - Portland, Portland, Oregon, United States